CLINICAL TRIAL: NCT04609644
Title: Digital Tools for Improved Awareness and Self-Management of Asthma in Adults
Brief Title: Asthma Digital Study
Acronym: ADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elevance Health (Industry)
Collaborators: Apple Inc. (Industry); University of California, Irvine (Other); HealthCore, Inc. (Industry); CareEvolution, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HS# 2020-5711
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Passive (No Intervention): Passive arm participants will be sent two devices, at no cost-an Apple Watch and a Beddit Sleep Monitor. These are commercially available and have not been modified for this study. Participants will be asked to use these devices regularly throughout study Year 1. Participants can optionally continue to use devices during Year 2, if they have met requirements during Year 1 to keep study devices. To be eligible to keep devices, participants must meet pre-specified levels of adherence to study procedures.
  Access to the Study App will be provided to all participants. It will be used to administer informed consent and electronic patient reported outcome (ePRO) measures, and for other study purposes. However, passive participants will not have access to the Study App features designed to support asthma self-management.
- Active (Experimental): Active arm participants will be sent the same devices, also at no cost, and asked to use them in the same manner.
  Only the active arm will have access to Study App features for asthma self-management, including:
  * "Smart nudges" that may promote proactive asthma self-management
  * Asthma symptom and trigger tracking
  * Evidence-based asthma education
  * The ability to photograph and easily reference an asthma action plan from a healthcare provider.
  * A 90-day summary of self-reported asthma symptoms/triggers and device-recorded heart rate and respiratory rate. This summary can be shared with providers.
  * In-app viewing of active asthma medications, refills available, and phone numbers to call for refills (subject to prescription benefits).
  Active participants can, but are not required to, use the Study App in Year 2. Those who choose to may keep using study devices in Year 2, provided they meet requirements to keep devices. These requirements are the same for both arms.
  Interventions: Other: Digital Tools for Asthma Self-Management

INTERVENTIONS:
Other: Digital Tools for Asthma Self-Management — Please see description of active study arm.
  Arms: Active

SUMMARY:
The Asthma Digital Study is a virtual, two-arm, randomized, controlled trial that will investigate the impact of digital tools on asthma symptom control, exacerbation frequency, healthcare utilization, and medical expenditures in adults with asthma.

DETAILED DESCRIPTION:
The Asthma Digital Study is a virtual, two-arm, randomized, controlled trial that will investigate the impact of digital tools on asthma symptom control, exacerbation frequency, healthcare utilization, and medical expenditures. Adults with asthma will be randomized to the passive or active arm in a 1:1 ratio.

All participants will be sent two devices, at no cost-an Apple Watch and a Beddit Sleep Monitor. These are publicly available, commercial devices that have not been modified for this study.

The study will be administered largely through a customized version of CareEvolution's MyDataHelps app (the "Study App"). Access to the Study App will be provided to all participants. It will be used to administer informed consent and electronic patient reported outcome (ePRO) measures, and for other study purposes. Only active arm participants will have access to Study App features designed to support asthma self-management. These features include "smart nudges" based on device data, symptom and trigger tracking, evidence-based education, summaries of health metrics gathered from the Apple Watch and Beddit Sleep Monitor, in-app medication refill resources, as well as other resources.

The study duration is 2 years. Participants can keep using the Study App and devices after Year 1, though this is not required. Primary analyses will utilize Year 1 data only. During Year 2, data collection will continue where available, though fewer data will be collected because use of digital tools is not required during Year 2, and health coverage changes may cause loss of access to claims data.

ELIGIBILITY:
Inclusion Criteria:

* Health insurance coverage through an Anthem, Inc. affiliate.
* 18-64 years of age
* Resident of the United States for the duration of the study
* Comfortable reading and writing in English
* Owns an iPhone 6s or later
* Has been diagnosed with asthma by a provider
* 1+ emergency department visit in the preceding 24 months with an associated asthma diagnosis, or a combination of factors that might be associated with uncontrolled asthma. Factors include:

  * History of asthma medication prescriptions
  * History of asthma-associated primary care visits
  * Diagnosis of chronic sinusitis, pharyngitis, influenza, allergic rhinitis, hypertension, diabetes, and/or obesity
  * History of smoking
  * Age and zip code

Exclusion Criteria:

* Unable to sleep in a bed with a Beddit sleep monitor at least 5 nights per week on average (e.g., shift workers who experience limited or erratic night-time sleep schedule, frequent travelers unable to stably sleep on the sensor at the requisite rate)
* Currently enrolled in any other asthma or pulmonary studies
* Currently on any immunologic for asthma
* Participated in a prior pilot study investigating the same digital tools
* Member of an Anthem plan with annual incentives limits of $100 or less
* Resident of Puerto Rico
* Pregnancy
* Diagnosis of any of the following:
* Chronic Obstructive Pulmonary Disease/Emphysema
* Cystic Fibrosis
* Any malignancy other than a non-melanoma skin cancer
* Any dementia diagnosis
* Neurodegenerative diseases (e.g., Parkinson's)
* Schizophrenia
* Heart failure
* On dialysis
* Women who are postpartum, with delivery in the past 8 weeks

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 901 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
Change in asthma-associated expenditures due to emergency department and hospital utilization | 12 months before and after baseline
  Sum of all allowed costs for emergency and hospital care, where asthma is specified as a diagnosis. Costs from the 12 months preceding baseline will be compared to costs from 12 months after baseline. Mean change in costs will be compared across arms.
Change from baseline in Asthma Control Test (ACT), a validated patient-reported outcome (PRO) measure of asthma symptom control | Baseline and 12-month time points
  ACT change among all participants with baseline ACT score suggesting that asthma may be uncontrolled (ACT score of 19 or lower). Mean ACT change will be compared across arms.

SECONDARY OUTCOMES:
Change from baseline in Asthma Control Test (ACT), a validated patient-reported outcome (PRO) measure of asthma symptom control | Active arm only: Baseline and months 1, 2, 3, 4, 5, 6, 8, 10, 12
  Change from baseline among active arm participants with baseline ACT score suggesting that asthma may be uncontrolled (ACT score of 19 or lower).
Adherence to Refills and Medications Scale, 7-item version (ARMS-7) | Active arm only: 2 weeks and months 2, 4, 6, 8, 10, 12
  Validated PRO measure of medication adherence
Readiness ruler, asthma self-management | Active arm only: 2 weeks and months 2, 4, 6, 8, 10, 12
  PRO measuring confidence in, and perceived importance of, asthma self-management
Work Productivity and Activity Impairment Questionnaire 2.0, asthma version | Active arm only: Baseline and months 1, 3, 5, 8, 12
  Validated PRO measure of asthma-associated work productivity impairment
Health Confidence Score | Active arm only: Baseline and months 1, 3, 5, 8, 12
  Validated PRO measure of confidence in ability to manage general health
Self-reported smoking and e-cigarette use | Baseline and month 12
  Adaptations of validated PRO measures
Symptom-free days | Active arm only: Months 1-12
  Measured using Study App
Frequency of prescriptions for oral corticosteroids | Months 1-12; Months 13-24
Asthma Medication Ratio | Months 1-12; Months 13-24
  For details see: www.ncqa.org/hedis/measures/medication-management-for-people-with-asthma-and-asthma-medication-ratio/
Adherence to asthma medications | Months 1-12; Months 13-24
  Proportion of days covered, measured using pharmacy claims
Asthma-associated expenditures due to emergency department and hospital utilization | Months 13-24
  Computed in the same manner as the primary outcome, except that expenditures are computed for Year 2 rather than Year 1.
Total Asthma-Associated Expenditures | Months 1-12; Months 13-24
  Total allowed costs for all care associated with asthma, including pharmacy and other costs
Total Medical Expenditures | Months 1-12; Months 13-24
  Total allowed costs for all claimed healthcare expenses
Frequency of unplanned visits for asthma care | Months 1-12; Months 13-24
  Includes acute primary care visits, urgent care visits, emergency visits
Study App Engagement Metrics | Active arm only: Months 1-12; Months 13-24
  Frequencies of symptom tracking, trigger tracking, app opens
Rates of enrollment in pharmacy auto-refill and home delivery services | Months 1-12; Months 13-24

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan Silberman, Palo Alto, California, United States

REFERENCES:
- [Background] Silberman J, Sarlati S, Harris B, Bokhari W, Boushey H, Chesnutt A, Zhu P, Sitts K, Taylor TH, Willey VJ, Fuentes E, LeKrey M, Hou E, Kaur M, Niyonkuru C, Muscioni G, Bianchi MT, Bota DA, Lee RA. A digital approach to asthma self-management in adults: Protocol for a pragmatic randomized controlled trial. Contemp Clin Trials. 2022 Nov;122:106902. doi: 10.1016/j.cct.2022.106902. Epub 2022 Aug 30. PMID 36049674
- [Background] Harris B, Silberman J, Sarlati S, et al. A digital asthma self-management tool reduced emergency visit rates in a Medicaid population. Ann Allergy Asthma Immunol. 2023;131(5):S230-S231. doi:10.1016/j.anai.2023.10.021
- [Derived] Silberman J, Sarlati S, Harris B, Lenyoun H, Kaur M, Wagner BG, Bokhari W, Boushey H, Chesnutt A, Sitts K, Zhu P, Willey VJ, Fuentes E, LeKrey M, Alger BL, Muscioni G, Bianchi MT, Bota DA, Taylor TH, Evans M, Amin AN, Stark D, Montanari C, Perry JS, Vian C, Patel M, Poe W, Lee RA. A Digital Asthma Self-Management Program for Adults: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2521438. doi: 10.1001/jamanetworkopen.2025.21438. PMID 40674052